CLINICAL TRIAL: NCT00054106
Title: A Phase I Study Of Combination Neoadjuvant Hormone Therapy And Weekly OGX-011 (Clusterin Antisense Oligonucleotide) Prior To Radical Prostatectomy In Patients With Localized Prostate Cancer
Brief Title: Hormone Therapy and OGX-011 Before Radical Prostatectomy in Treating Patients With Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I153; CAN-NCIC-IND153 (Other: PDQ); ONCOGENEX-OGX-01-01 (Other: Oncogenex Technologies); CDR0000269888 (Other: PDQ)
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2020-04

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage III prostate cancer; stage II prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Buserelin; Flutamide; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: buserelin
Drug: custirsen sodium
Drug: flutamide
Procedure: conventional surgery
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Androgens can stimulate the growth of prostate cancer cells. Drugs such as flutamide and buserelin may stop the adrenal glands from producing androgens. OGX-011 may help flutamide and buserelin kill more tumor cells by making tumor cells more sensitive to the drugs. Giving flutamide and buserelin with OGX-011 before surgery may shrink the tumor so it can be removed during surgery.

PURPOSE: Phase I trial to study the effectiveness of combining hormone therapy with OGX-011 before radical prostatectomy in treating patients who have prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose and recommended phase II dose of OGX-011 (clusterin antisense oligonucleotide) when administered with neoadjuvant hormonal therapy before radical prostatectomy in patients with adenocarcinoma of the prostate.
* Determine the toxicity of this regimen in these patients.
* Determine the pharmacokinetics of OGX-011 when this regimen is administered in these patients..
* Assess the effects of this regimen on pathologic complete response rates in these patients.
* Correlate plasma and/or prostate concentrations of OGX-011 with patient response or toxicity measures.

OUTLINE: This is a dose-escalation study of OGX-011.

Patients receive OGX-011 IV over 2 hours on days 1, 3, 5, 8, 15, 22, and 29; oral flutamide three times daily for 4 weeks; and buserelin subcutaneously on day 1.

Cohorts of 3-6 patients (except for 1 patient at starting dose) receive escalating doses of OGX-011 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. The recommended phase II dose is the dose preceding the MTD.

Patients undergo radical prostatectomy and bilateral pelvic lymphadenectomy 1 week after the last dose of neoadjuvant therapy.

Patients are followed at 7 days after surgery and then at 3 months.

PROJECTED ACCRUAL: Approximately 25-33 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate

  * High-risk, localized disease that is previously untreated
  * Minimum of 2 positive biopsies
  * Meets at least 1 of the following criteria:

    * Stage T3
    * Serum PSA greater than 10 ng/mL
    * Gleason score 7-10
    * Gleason score 6 and at least 3 positive biopsies
* Potential candidate for radical prostatectomy

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* WBC at least 3,000/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10.0 g/dL

Hepatic

* Bilirubin normal
* AST and ALT normal
* PTT normal
* INR normal

Renal

* Creatinine normal

Cardiovascular

* No significant cardiac dysfunction

Other

* Fertile patients must use effective contraception
* No known hypersensitivity to oligonucleotides, luteinizing hormone-releasing hormone analogs, or anti-androgens
* No evidence of active uncontrolled infection
* No other malignancy within the past 5 years except adequately treated nonmelanoma skin cancer
* No other serious illness, psychiatric disorder, or medical condition that would preclude study compliance
* No history of a significant neurological disorder that would preclude informed consent
* No geographical condition that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy for prostate cancer

Endocrine therapy

* No prior hormonal therapy for prostate cancer

Radiotherapy

* No prior radiotherapy for prostate cancer
* No concurrent radiotherapy

Surgery

* Not specified

Other

* No concurrent heparin or warfarin anticoagulation
* No other concurrent investigational therapy
* No other concurrent cytotoxic therapy

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2002-12-10 (Actual); Primary Completion 2004-09-23 (Actual); Study Completion 2008-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kim N. Chi, MD, Study Chair — British Columbia Cancer Agency
Locations (1):
- British Columbia Cancer Agency - Vancouver Cancer Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chi KN, Eisenhauer E, Fazli L, Jones EC, Goldenberg SL, Powers J, Tu D, Gleave ME. A phase I pharmacokinetic and pharmacodynamic study of OGX-011, a 2'-methoxyethyl antisense oligonucleotide to clusterin, in patients with localized prostate cancer. J Natl Cancer Inst. 2005 Sep 7;97(17):1287-96. doi: 10.1093/jnci/dji252. PMID 16145049
- [Result] Chi KN, Eisenhauer E, Fazli L, et al.: A phase I pharmacokinetic (PK) and pharmacodynamic (PD) study of OGX-011, a 2'methoxyethyl phosphorothioate antisense to clusterin, in patients with prostate cancer prior to radical prostatectomy. [Abstract] J Clin Oncol 22 (Suppl 14): A-3033, 203s, 2004.